CLINICAL TRIAL: NCT00949728
Title: Conjunctival Autologous Transplantation Using Fibrin Glue in Primary Pterygia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Olhos Sadalla Amin Ghanem (Other)
Responsible Party: Ramon Coral Ghanem, Sadalla Amin Ghanem Eye Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: cola106
Record Dates: First submitted 2009-07-17; First posted 2009-07-30 (Estimated); Last update posted 2009-07-30 (Estimated); Status verified 2009-07

CONDITIONS: Pterygium; Primary
Keywords: Pterygium; Autologous Transplantation; Conjunctiva; Fibrin Tissue Adhesive; Recurrence
MeSH Terms: conditions — Pterygium; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fibrin glue (Other)
  Interventions: Procedure: Conjunctival autograft using fibrin glue

INTERVENTIONS:
Procedure: Conjunctival autograft using fibrin glue — Conjunctival autograft using fibrin glue in pterygium surgery
  Other Names: Pterygium surgery using fibrin glue

SUMMARY:
To evaluate the recurrence and postoperative complications rates after conjunctival autograft surgery using fibrin adhesive for primary pterygium

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of primary pterygium
* Symptomatic pterygium
* Limbal invasion

Exclusion Criteria:

* Secondary pterygium

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2006-10; Primary Completion 2008-08 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Recurrence of pterygium after its excision with the conjunctival autograft technique. | One, three and five months after surgery.

SECONDARY OUTCOMES:
Postoperative complications following the pterygium excision, such as partial graft detachment, dellen, granuloma or sutures failure. | One day, one week and one month after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Renan F Oliveira, Principal Investigator; Ramon C Ghanem, M.D., Study Director — Sadalla Amin Ghanem Eye Hospital
Locations (1):
- Sadalla Amin Ghanem Eye Hospital, Joinville, Santa Catarina, Brazil

REFERENCES:
- [Background] Koranyi G, Seregard S, Kopp ED. Cut and paste: a no suture, small incision approach to pterygium surgery. Br J Ophthalmol. 2004 Jul;88(7):911-4. doi: 10.1136/bjo.2003.032854. PMID 15205236
- [Background] Bahar I, Weinberger D, Gaton DD, Avisar R. Fibrin glue versus vicryl sutures for primary conjunctival closure in pterygium surgery: long-term results. Curr Eye Res. 2007 May;32(5):399-405. doi: 10.1080/02713680701294723. PMID 17514524
- [Background] Marticorena J, Rodriguez-Ares MT, Tourino R, Mera P, Valladares MJ, Martinez-de-la-Casa JM, Benitez-del-Castillo JM. Pterygium surgery: conjunctival autograft using a fibrin adhesive. Cornea. 2006 Jan;25(1):34-6. doi: 10.1097/01.ico.0000164780.25914.0a. PMID 16331038